CLINICAL TRIAL: NCT04667221
Title: Cognitive Improvement Through Transcranial Direct Current Stimulation for Patients With Multiple Sclerosis
Brief Title: Cognitive Improvement Through tDCS for Patients With Multiple Sclerosis
Acronym: MS-CICS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: MS-CICS
Record Dates: First submitted 2020-12-08; First posted 2020-12-14 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Randomized, balanced crossover design.
Who Masked: Participant, Investigator
Masking Description: Participants and investigators are blinded according to the sham / active stimulation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Anodal transcranial direct current stimulation (Experimental): Patients will be bilaterally stimulated with anodal tDCS at the parietal cortex (Brodmann Area 7).
  Interventions: Device: Active transcranial direct current stimulation
- Cathodal transcranial direct current stimulation (Experimental): Patients will be bilaterally stimulated with cathodal tDCS at the parietal cortex (Brodmann Area 7).
  Interventions: Device: Active transcranial direct current stimulation
- Sham transcranial direct current stimulation for anodal group (Sham Comparator): Patients will be bilaterally stimulated with sham tDCS at the parietal cortex (Brodmann Area 7). As a consequence of the crossover design, both experimental arms receive sham stimulation.
  Interventions: Device: Sham transcranial direct current stimulation
- Sham transcranial direct current stimulation for cathodal group (Sham Comparator): Patients will be bilaterally stimulated with sham tDCS at the parietal cortex (Brodmann Area 7). As a consequence of the crossover design, both experimental arms receive sham stimulation.
  Interventions: Device: Sham transcranial direct current stimulation

INTERVENTIONS:
Device: Active transcranial direct current stimulation — A high-definition tDCS set-up will be used with a battery-driven stimulator (Starstim 8, Neuroelectrics). Active stimulation will be conducted with 1.5 milliampere (mA) with two electrodes using three reference electrodes for each active one for 20 minutes.
  Other Names: non-invasive brain stimulation; transcranial electrical stimulation
  Arms: Anodal transcranial direct current stimulation; Cathodal transcranial direct current stimulation
Device: Sham transcranial direct current stimulation — A high-definition tDCS set-up will be used with a battery-driven stimulator (Starstim 8, Neuroelectrics). Sham stimulation will have a 40 seconds ramp-up and down. No stimulation will be applied after this 40 seconds.
  Other Names: non-invasive brain stimulation; transcranial electrical stimulation
  Arms: Sham transcranial direct current stimulation for anodal group; Sham transcranial direct current stimulation for cathodal group

SUMMARY:
Multiple sclerosis (MS) is a chronic inflammatory disease with around 200.000 patients in Germany. Besides physical symptoms, cognitive resources degrade over the years. Transcranial direct current stimulation (tDCS) is an established procedure to modulate cortical excitability in motor and cognitive functions. Therefore, tDCS may improve cognitive functions in patients with MS. Patients will work on a modified version of the symbol digits modalities test in two experimental sessions. During the task, they will receive either active stimulation or sham stimulation in a crossover design. Active stimulation is divided in anodal and cathodal stimulation. Anodal stimulation should facilitate cognitive processing; cathodal stimulation, on the other hand, should hinder cognitive processing.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a chronic inflammatory autoimmune disease characterized by a multitude of symptoms, which greatly reduce the quality of life of patients. In addition to sensory and visual sensory disorders, movement disorders, paresis, fatigue and other physical symptoms, 65-95% of patients with MS also suffer from cognitive impairments. These cognitive impairments develop in the later course of the disease and express themselves in slower processing speed, delays in learning and memory performance, and executive dysfunction. In recent years, non-pharmacological approaches aimed at improving cognitive performance in MS have increasingly come into focus, including the transcranial direct current stimulation (tDCS).

TDCS has only been investigated in a few studies that had the aim to improve cognitive performance in MS. Further, it has only been carried out in combination with cognitive training paradigms and repeated stimulation sessions. Mattioli and colleagues (2016) could e.g. show that after 10 sessions of cognitive training with tDCS stimulation of the dorsolateral prefrontal cortex, there was greater improvement in symbol-digit modalities test (SDMT) in the experimental group than in the control group. Similarly, Charvet and colleagues (2018) showed that after 10 sessions of cognitive training with simultaneous tDCS stimulation of the dorsolateral prefrontal cortex, the experimental group showed a significant improvement in the domains of attention and response variability compared to the control group. These studies therefore reflect an interaction between cognitive training and tDCS, and do not allow any conclusions to be drawn about the effect of tDCS on specific processes. It is not yet known whether tDCS alone can positively influence specific cognitive functional impairments.

Therefore, the present study wants to investigate whether acute application of tDCS can improve specific cognitive functions. An adapted version of the clinically SDMT was conducted, as this test is one of the most widely used tests to describe cognitive impairments in MS. Based on a meta-analysis by Silva and colleagues (2018), that shows which brain areas are related to the implementation of the SDMT, the parietal cortex (BA7) is stimulated bilaterally with either excitatory (anodal) or inhibitory (cathodal) tDCS.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of multiple sclerosis.
* no acute inflammation during the last 3 months before the experimental intervention.
* no cortisol treatment during the last 3 months before the experimental intervention.
* stable medication during the experimental intervention.
* unrestrained or corrected visual ability.
* ability to read and write short german sentences.
* adequate motor ability to give responses on a keyboard.
* German as main language.

Exclusion Criteria:

* major depressive symptoms or any further neurological and/or psychiatric disease at experimental intervention.
* standard tDCS exclusion criteria (e.g. cardiac pacemaker, metal implants in head region, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-12-08 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Reaction Times in symbol-digit modalities test. | Assessed at two timepoints (1x during active (anodal/cathodal) tDCS intervention at Day 1 or 7 (depends on randomization), 1x during sham tDCS intervention at Day 1 or 7 (depends on randomization))
  Reaction times in milliseconds for the performance of the symbol-digit modalities test.

SECONDARY OUTCOMES:
Hit Rate in symbol-digit modalities test. | Assessed at two timepoints (1x during active (anodal/cathodal) tDCS intervention at Day 1 or 7 (depends on randomization), 1x during sham tDCS intervention at Day 1 or 7 (depends on randomization))
  Hit rate in percentage of correct responses in the symbol-digit modalities test.
Baseline performance in symbol-digit modalities test. | Assessment at baseline (Day 0, before stimulation).
  Baseline performance of paper-pencil version of the symbol-digit modalities test as a predictor for the stimulation effect.

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Meinzer, Prof., PhD, Principal Investigator — Universitymedicine Greifswald
Locations (1):
- University Medicine Greifswald, Greifswald, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Riemann S, Mittelstadt M, Glatzki M, Zilges C, Wolff C, Niemann F, Roheger M, Floel A, Grothe M, Meinzer M. Information processing speed modulation by electrical brain stimulation in multiple sclerosis: towards individually tailored protocols. Brain Commun. 2025 Jun 6;7(3):fcaf223. doi: 10.1093/braincomms/fcaf223. eCollection 2025. PMID 40574976